CLINICAL TRIAL: NCT04684043
Title: Prognostic Implications of Physiologic Investigation After Revascularization With Stent
Acronym: POST-PCI FLOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bon-Kwon Koo (Other)
Collaborators: Inje University Ilsan Paik Hospital, Goyang, South Korea (Unknown); Nanjing First Hospital, Nanjing Medical University, Nanjing, China (Unknown); Tsuchiura Kyodo General Hospital (Other); McGovern Medical School at UTHealth and Memorial Hermann Hospital, TX, USA (Unknown); Nagoya City University Graduate School of Medical Science, Nagoya, Japan (Unknown); Rutgers Robert Wood Johnson Medical School (Other); Cardiovascular Center Aalst, OLV Clinic, Aalst, Belgium (Unknown); San Raffaele Scientific Institute, Milan, Italy (Unknown); Ajou University Hospital, Suwon, South Korea (Unknown); University of Cincinnati (Other); Kyoto Second Red Cross Hospital, Kyoto, Japan (Unknown); Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Korea (Unknown); Tokyo Medical University Hachioji Medical Center, Tokyo, Japan (Unknown)
Responsible Party: Sponsor-Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: H-2009-042-1155
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Coronary Disease
Keywords: fractional flow reserve; percutaneous coronary intervention; drug-eluting stent; coronary atherosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post PCI state: The study population of this study underwent percutaneous coronary intervention(PCI) with drug-eluting stent (DES) and measured fractional flow reserve after PCI.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI was performed using drug-eluting stents

SUMMARY:
Percutaneous coronary intervention (PCI) is a standard treatment strategy for coronary artery disease (CAD). With the presence of myocardial ischemia, PCI reduces the risks of death, myocardial infarction (MI) and revascularization compared to medical therapy. However, the risk of future clinical events remains high, and about 10% of patients experienced further cardiovascular events after PCI. Several factors are associated with these poor outcomes. Well known patient-related risk factors are diabetes mellitus, chronic kidney disease, left ventricular dysfunction, previous MI, and presentation with the acute coronary syndrome. Procedure-related factors, such as stent underexpension, malapposition, edge dissection, the number of the used stent, and total stent length, are also related to poor prognosis after PCI. Recent studies reported that fractional flow reserve (FFR) after coronary stenting, or post PCI FFR, was associated with future clinical outcomes after PCI, and low post PCI FFR value was associated with procedural factors. However, optimal cut-off values of post-PCI FFR ranged widely, from 0.86 to 0.96, and some study reported the limited prognostic value of post-PCI FFR. This might result from differences in study populations, the definition of outcomes, type of stent used, and distribution of included vessels among previous studies.

To establish the clinical relevance of post-PCI FFR and to evaluate the useful cut-off value of post-PCI FFR in daily practice, investigators planned to incorporate all previous evidence of post-PCI FFR by collaboration with international researchers.

DETAILED DESCRIPTION:
This study population was incorporated from studies which were already published. Investigators will incorporate all known registries to the POST-PCI FLOW registry by requesting data from principal investigator of each registry.

Investigators will perform systemic review of the previous published data and an updated patient-level meta-analysis of studies, including the most recent publications. PubMed, EMBASE, Cochrane Central Register of Controlled Trials, the United States National Institutes of Health registry of clinical trials, and relevant websites were searched for pertinent published studies. The electronic search strategy was complemented by manual examination of references cited by included articles, recent reviews, editorials, and meta-analyses. No restrictions were imposed on language, study period, or sample size. Searching key words included 'post', 'after', 'PCI', 'Percutaneous coronary intervention', 'coronary stenting', 'stenting', 'stent', 'stent implantation', 'FFR', and 'fractional flow reserve'.

ELIGIBILITY:
Articles were included when they met the following prespecified criteria: (1) included the patients who underwent PCI with drug-eluting stent (DES); (2) post-PCI FFR was measured after DES implantation; (3) pre-PCI FFR measurement was not mandatory for article inclusion; (4) patients were followed up at least 6 months; (5) clinical outcomes, including all-cause death, cardiac death, target vessel myocardial infarction (TVMI) or target vessel revascularization (TVR), were clearly reported; (6) randomized controlled trials or non-randomized prospective or retrospective registries were included. Two independent investigators screened titles and abstracts, identified duplicated studies, performed full-article reviews, and determined the studies' inclusion. The third investigator supervised the searching process and adjudicated all the disagreements.

* Patients with life expectancy < 2 years.

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as obstructive coronary artery disease and treated by DES and measured post PCI FFR after PCI.
Sampling Method: Non-Probability Sample
Enrollment: 5100 (Estimated)
Dates: Start 2020-05-16 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 2 years
  A composite of cardiac death, target vessel myocardial infarction and target vessel revascularization

SECONDARY OUTCOMES:
Cardiac death or myocardial infarction | 2 years
  a composite of cardiac death and target vessel myocardial infarction
Target vessel myocardial infarction | 2 years
Target vessel revascularization | 2 years

OTHER OUTCOMES:
Cut-off value of post-PCI FFR | 2 years
  Define the best cut-off value for predicting the future adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — Seoul National University Hospital, Seoul, South Korea; Joon Hyung MD, PhD, MD, PhD, Principal Investigator — Inje University Ilsan Paik Hospital, Goyang, South Korea; Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University, Nanjing, China; Tsunekazu Kakuta, MD, PhD, Principal Investigator — Tsuchiura Kyodo General Hospital; Nils P. Johnson, MD, MS, Principal Investigator — McGovern Medical School at UTHealth and Memorial Hermann Hospital, TX, USA; Tsuyoshi Ito, MD, Principal Investigator — Nagoya City University Graduate School of Medical Science, Nagoya, Japan; Abdul Hakeem, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School; Bernard De Bruyne, MD, PhD, Principal Investigator — Cardiovascular Center Aalst, OLV Clinic, Aalst, Belgium; Lorenzo Azzalini, MD, PhD, Principal Investigator — San Raffaele Scientific Institute, Milan, Italy; Hong-Seok Lim, MD, PhD, Principal Investigator — Ajou University Hospital, Suwon, South Korea; Massoud A. Leesar, MD, PhD, MSc, Principal Investigator — University of Cincinnati; Akiko Matsuo, MD, Principal Investigator — Kyoto Second Red Cross Hospital, Kyoto, Japan; Nobuhiro Tanaka, MD, PhD, MSc, Principal Investigator — Tokyo Medical University Hachioji Medical Center, Tokyo, Japan; Joo Myung Lee, MD, PhD, MSc, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, Select, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Fearon WF, Nishi T, De Bruyne B, Boothroyd DB, Barbato E, Tonino P, Juni P, Pijls NHJ, Hlatky MA; FAME 2 Trial Investigators. Clinical Outcomes and Cost-Effectiveness of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease: Three-Year Follow-Up of the FAME 2 Trial (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation). Circulation. 2018 Jan 30;137(5):480-487. doi: 10.1161/CIRCULATIONAHA.117.031907. Epub 2017 Nov 2. PMID 29097450
- [Background] Hwang D, Lee JM, Lee HJ, Kim SH, Nam CW, Hahn JY, Shin ES, Matsuo A, Tanaka N, Matsuo H, Lee SY, Doh JH, Koo BK. Influence of target vessel on prognostic relevance of fractional flow reserve after coronary stenting. EuroIntervention. 2019 Aug 29;15(5):457-464. doi: 10.4244/EIJ-D-18-00913. PMID 30561367
- [Background] Li SJ, Ge Z, Kan J, Zhang JJ, Ye F, Kwan TW, Santoso T, Yang S, Sheiban I, Qian XS, Tian NL, Rab TS, Tao L, Chen SL. Cutoff Value and Long-Term Prediction of Clinical Events by FFR Measured Immediately After Implantation of a Drug-Eluting Stent in Patients With Coronary Artery Disease: 1- to 3-Year Results From the DKCRUSH VII Registry Study. JACC Cardiovasc Interv. 2017 May 22;10(10):986-995. doi: 10.1016/j.jcin.2017.02.012. Epub 2017 Apr 26. PMID 28456699
- [Background] Rimac G, Fearon WF, De Bruyne B, Ikeno F, Matsuo H, Piroth Z, Costerousse O, Bertrand OF. Clinical value of post-percutaneous coronary intervention fractional flow reserve value: A systematic review and meta-analysis. Am Heart J. 2017 Jan;183:1-9. doi: 10.1016/j.ahj.2016.10.005. Epub 2016 Oct 11. PMID 27979031
- [Background] van Zandvoort LJC, Masdjedi K, Witberg K, Ligthart J, Tovar Forero MN, Diletti R, Lemmert ME, Wilschut J, de Jaegere PPT, Boersma E, Zijlstra F, Van Mieghem NM, Daemen J. Explanation of Postprocedural Fractional Flow Reserve Below 0.85. Circ Cardiovasc Interv. 2019 Feb;12(2):e007030. doi: 10.1161/CIRCINTERVENTIONS.118.007030. PMID 30732469
- [Derived] Choi KH, Kwon W, Shin D, Lee SH, Hwang D, Zhang J, Nam CW, Shin ES, Doh JH, Chen SL, Kakuta T, Toth GG, Piroth Z, Hakeem A, Uretsky BF, Hokama Y, Tanaka N, Lim HS, Ito T, Matsuo A, Azzalini L, Leesar MA, Daemen J, Collison D, Collet C, De Bruyne B, Koo BK, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Differential Impact of Fractional Flow Reserve Measured After Coronary Stent Implantation by Left Ventricular Dysfunction. JACC Asia. 2023 Dec 12;4(3):229-240. doi: 10.1016/j.jacasi.2023.10.009. eCollection 2024 Mar. PMID 38463680
- [Derived] Yang S, Hwang D, Zhang J, Park J, Yun JP, Lee JM, Nam CW, Shin ES, Doh JH, Chen SL, Kakuta T, Toth GG, Piroth Z, Johnson NP, Hakeem A, Uretsky BF, Hokama Y, Tanaka N, Lim HS, Ito T, Matsuo A, Azzalini L, Leesar MA, Neleman T, van Mieghem NM, Diletti R, Daemen J, Collison D, Collet C, De Bruyne B, Koo BK. Clinical and Vessel Characteristics Associated With Hard Outcomes After PCI and Their Combined Prognostic Implications. J Am Heart Assoc. 2023 Sep 5;12(17):e030572. doi: 10.1161/JAHA.123.030572. Epub 2023 Aug 29. PMID 37642032